CLINICAL TRIAL: NCT05943782
Title: Functional Evaluation of CAD/CAM Onlays Fabricated by Subtractive Versus Additive Digital Manufacturing Techniques. A One Year Randomized Clinical Trial.
Brief Title: Evaluation of CAD/CAM Onlays Fabricated by Subtractive Versus Additive Digital Manufacturing Techniques.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 052308
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-05

CONDITIONS: Caries,Dental; Broken Teeth; Fracture Tooth; Defective Dentition
MeSH Terms: conditions — Dental Caries; Tooth Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- additive manufacturing of onlays (Experimental): additive CAD/CAM manufacturing of dental restorations by 3D printing
  Interventions: Procedure: Onlay manufactured by 3D printing
- subtractive manufacturing of onlays (Active Comparator): subtractive CAD/CAM manufacturing of dental restorations by milling
  Interventions: Procedure: onlay manufactured by milling

INTERVENTIONS:
Procedure: onlay manufactured by milling — indirect restorations for treating mutilated molars manufactured by CAD/CAM subtractive technique
  Arms: subtractive manufacturing of onlays
Procedure: Onlay manufactured by 3D printing — indirect restorations for treating mutilated molars manufactured by CAD/CAM additive technique
  Arms: additive manufacturing of onlays

SUMMARY:
Aim of the study: The aim of this RCT is to evaluate CAD/CAM onlays fabricated by subtractive technique (brilliant crios) versus additive technique (varseosmile crown plus material), in terms of clinical functional evaluation following the FDI criteria and three-dimensional digital evaluation of the marginal and internal fit by triple scan protocol.

Materials and methods: A total of 30 patients will be enrolled in the clinical trial following the eligibility criteria. Then, the patients will be randomly allocated to receive either 3D printed onlays or milled ones. A blinded operator will prepare a standardized cavity for the restoration and an impression will be performed. After designing the restoration on the Exocad software, A dentist not involved in the clinical part of the study will receive the STL file of the design and envelopes containing the information necessary only to manufacture the restorations (tooth numbers and restorative materials) to proceed with either the milling or printing procedures. Try in and cementation procedures will be similarly performed for both groups by a blinded operator. Finally, the marginal and internal fit will be evaluated by using the triple scan protocol for digital 3D assessment.

Also, a baseline, six months and 12 months assessments will be performed by a blinded examiner, not involved in the clinical part for assessing the functional clinical performance of the re3stprations using the FDI criteria. Finally, the data will be statistically analyzed.

DETAILED DESCRIPTION:
Statement of the problem: Several randomized clinical trials (RCT) investigated the clinical performance of milled ceramic and composite posterior indirect adhesive restorations. However, none investigated that of 3D printed ones and the differences in their fabrication process and material properties of these restorations may impact their clinical performance. Therefore, clinical assessment of that novel additive technique is required.

Aim of the study: The aim of this RCT is to evaluate CAD/CAM onlays fabricated by subtractive technique (brilliant crios) versus additive technique (varseosmile crown plus material), in terms of clinical functional evaluation following the FDI criteria and three-dimensional digital evaluation of the marginal and internal fit by triple scan protocol.

Materials and methods: A total of 30 patients will be enrolled in the clinical trial following the eligibility criteria. Then, the patients will be randomly allocated to receive either 3D printed onlays or milled ones. A blinded operator will prepare a standardized cavity for the restoration and an impression will be performed. After designing the restoration on the Exocad software, A dentist not involved in the clinical part of the study will receive the STL file of the design and envelopes containing the information necessary only to manufacture the restorations (tooth numbers and restorative materials) to proceed with either the milling or printing procedures. Try in and cementation procedures will be similarly performed for both groups by a blinded operator. Finally, the marginal and internal fit will be evaluated by using the triple scan protocol for digital 3D assessment.

Also, a baseline, six months and 12 months assessments will be performed by a blinded examiner, not involved in the clinical part for assessing the functional clinical performance of the re3stprations using the FDI criteria. Finally, the data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of caries lesion, defective amalgam, or composite restorations in posterior dentition (molars), suitable for the restoration with ceramic onlays.
2. Presence of antagonist tooth.
3. Adult patients (age: 18-50 years) of both genders.
4. Good general and oral health; Able to tolerate necessary restorative procedures and willing to sign an informed consent.
5. Absence of orthodontic appliances.
6. Absence of malocclusion and tooth malformation.

Exclusion Criteria:

1. Presence of non-carious cervical lesions.
2. Pregnant women.
3. Allergy to any of the restorative materials.
4. Mobile teeth, indicating periodontal disease or trauma.
5. External or internal resorption.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Marginal and internal fit. | Immediate after treatment
  three-dimensional digital evaluation by triple scan protocol in microns

SECONDARY OUTCOMES:
clinical functional evaluation . | one year
  clinical functional evaluation following the FDI criteria by clinical examination performed by trained investigators

IPD SHARING:
Plan to Share IPD: No